CLINICAL TRIAL: NCT04226677
Title: Investigation of the Effects of Video Based Training and Aerobic Exercise Training on Game Addiction Level and Functional Performance in Individuals With Internet Gaming Disorder
Brief Title: The Effects of Video Based Training and Aerobic Exercise Training in Individuals With Internet Gaming Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cagtay Maden (Other)
Responsible Party: Sponsor-Investigator, Cagtay Maden, research assistant,physiotherapist, Hasan Kalyoncu University
Organization: Hasan Kalyoncu University (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/111
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Gaming Disorder; Sedentary Behavior
Keywords: gaming disorder; aerobic exercise; exergame
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise; Exergaming; Control Groups

STUDY DESIGN:
Intervention Model Description: participants are grouped randomly, the first group is the aerobic exercise group, the second group is the video based exercise group and the third group is the combination of these.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aerobic exercise group (Experimental): Aerobic exercise group is received treadmill training.
  Interventions: Other: aerobic exercise
- Video based exercise group (Experimental): Video based exercise group is received exergame training.
  Interventions: Other: Video based exercise
- Control group (Experimental): Control group
  Interventions: Other: Control group

INTERVENTIONS:
Other: aerobic exercise — Treadmill training is include warming, cooling and training phase according to rating of perceived exertion for participants.
  Other Names: Treadmill training
  Arms: aerobic exercise group
Other: Video based exercise — Exergame training include virtual reality games by xbox kinect.
  Other Names: exergame
  Arms: Video based exercise group
Other: Control group — first and last evaluations will be made
  Other Names: no intervention
  Arms: Control group

SUMMARY:
In this study, video-based training, aerobic training and both training will be applied to individuals with internet gaming disorder. Addiction levels and functional performance will be evaluated before and after treatment.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of game-based training and aerobic exercise training on game addiction level, functional performance and exercise capacity in individuals with internet play disorder. In addition, the investigators think that facilitate the transition to exercise by using game-based training in order to gain exercise habit and reduce sedentary behaviours in individuals with internet gaming disorder.

ELIGIBILITY:
Inclusion Criteria:

* DSM V (Diagnostic and Statistical Manual of Mental Disorders, revision 5) Internet Gaming Impairment (IOOB) Diagnostic criteria: approval of five to nine items
* No communication barrier
* Playing game (smart phone,Play Station 4, Xbox, Personal Computer) at least 2 hours a day in the last year

Exclusion Criteria:

* Cigarette use over 10 packsXyear
* be using any medicine
* Be actively involved in any sport.
* Having chronic disease
* Having physical disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Internet Gaming Disorder Scale-Short-Form (IGDS9-SF) | 2 Monthly change
  It consists of 9 questions. The scores that can be obtained from the scale vary between 9 and 45 and the increase in the scores, especially 36 points and above, indicates the high risk of game addiction.
The International Physical Activity Questionnaire (IPAQ) | 2 Monthly change
  Used to calculate weekly physical activity level and METs

SECONDARY OUTCOMES:
Quality of Life Assessment: Short Form-36. | 2 Monthly change
  Short Form-36., quality of life questionnaire will be used. This questionnaire consists of questions measuring physical function, physical role limitation, pain, general health, vitality, social function, emotional role limitations, and mental health status. The scores that can be obtained from the scale vary between 0 and 100 and the increase in the scores indicates that the quality of life is high.
Anxiety Scale | 2 Monthly change
  Beck Anxiety Scale will be used to determine the anxiety levels of individuals.The scores that can be obtained from the scale vary between 0 and 30 and the increase in the scores indicates that the anxiety is high.
Senior Fitness Test (SFT) | 2 Monthly change
  It is a test with seven physical fitness test parameters. Time and length measurements are saved in these parameters.
20m-Shuttle Run Test | 2 Monthly change
  It is used to assess aerobic capacity with the treadmill. The maximum oxygen consumption is saved.

CONTACTS AND LOCATIONS:
Overall Officials: Çağtay maden, MSc, Pt, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu Universty, Gaziantep, Şahinbey, Turkey (Türkiye)